CLINICAL TRIAL: NCT01979289
Title: Computerized Cognitive Remediation for Geriatric Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K23MH095830 (NIH)
Record Dates: First submitted 2013-10-25; First posted 2013-11-08 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Major Depressive Disorder; Major Depressive Episode
Keywords: Executive Dysfunction; Cognitive Remediation; Geriatric; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Computer Treatment: Active (Experimental): Computerized Cognitive Remediation: Targeted to underlying cerebral networks associated with remission.
  Interventions: Other: computerized cognitive remediation
- Computer Treatment: Control (Active Comparator): Computerized Cognitive Remediation: Non-targeted
  Interventions: Other: computerized cognitive remediation:Control

INTERVENTIONS:
Other: computerized cognitive remediation
  Arms: Computer Treatment: Active
Other: computerized cognitive remediation:Control
  Arms: Computer Treatment: Control

SUMMARY:
This research study will examine if a targeted computerized cognitive remediation (CCR) training program is better for treating geriatric depression than general computer activity. We will also examine whether this intervention is related to improvement in cognitive and depressive symptoms. Elderly patients with depression, who have, and who have not been treated with antidepressant medication for their illness, will be recruited to participate in either a 30 hour cognitive remediation program or general computer activity designed to be both challenging and interesting. They will be asked to complete between 1 and 3 hours of remediation per day over 4 weeks. While undergoing the cognitive remediation participants will be asked questions to assess their symptoms of, as well as the severity of, their depression weekly. This will inform researchers about whether or not the CCR is helping to improve depressive symptoms. At the end of the CCR study, participants will be given a battery of cognitive tests design to tell investigators whether or not the CCR improved their thinking in a variety of different ways including improving attention, memory, and organization. Investigators will also determine whether changes in participants' thinking are related to changes in their mood or other depressive symptoms. It is hoped that information gained from this study will help investigators to better understand the brain processes associated with depression, recovery from depression, and will help inform the development of future alternative treatments for this illness.

ELIGIBILITY:
Inclusion Criteria:

Medicated Depressed Participants' Inclusion Criteria

1. Age: 60-89 years
2. Diagnosis: Major depression, unipolar (by DSM-IV criteria);
3. Severity of depression: MADRS >or =15 following at least 8-weeks of controlled antidepressant treatment.
4. No plans to change current antidepressant treatment.

Non-Medicated Depressed Participants' Inclusion Criteria

1. Age: 60-89 years
2. Diagnosis: Major depression, unipolar (by DSM-IV criteria);
3. Severity of depression: MADRS >or =15
4. No antidepressant treatment within the current episode. -

Exclusion Criteria:

1. Psychotic depression by DSM-IV, i.e., presence of delusions with a score higher than 2 (questionable delusion) rated by the Scale for Assessment of Positive Symptoms (SAPS) [47];
2. High suicide risk, i.e. intent or plan to attempt suicide in near future;
3. Presence of any Axis I psychiatric disorder (other than unipolar major depression) or substance abuse; Axis II diagnosis of antisocial personality (by SCID-P and DSM-IV);
4. History of psychiatric disorders other than unipolar major depression or generalized anxiety disorder (bipolar disorder, hypomania, and dysthymia are exclusion criteria);
5. Dementia: Mattis Dementia Rating Scale scores below 130 or diagnosis of dementia by DSM-IV; multiple sclerosis, history of head trauma or history of electroconvulsive therapy;
6. Amnestic Mild Cognitive Impairment (a-MCI), or Multiple Domain Mild Cognitive Impairment (md-MCI);
7. Acute or severe medical illness, i.e., delirium, metastatic cancer, decompensated cardiac, liver or kidney failure, major surgery, stroke or myocardial infarction during the three months prior to entry; or drugs known to cause depression, e.g., reserpine, alpha-methyl-dopa, steroids, sympathomimetics withdrawal;
8. Presence of a neurological brain disease and/or history of electroconvulsive therapy;
9. Current involvement in psychotherapy;
10. Inability to perform any of the ADLs (MAI: ADL subscale) even with assistance, e.g. walking with a cane is not an exclusion criterion;
11. Inability to speak English;
12. Aphasia;
13. Corrected visual acuity < 20/70; Color blindness -

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-08; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale | 4-6 weeks
  10 item measure to assess the core symptoms and cognitive features of clinical depression

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Shizuko Morimoto, Psy.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, White Plains, New York, United States